CLINICAL TRIAL: NCT01201876
Title: Reasons for Replacement or Repair of Dental Restorations
Brief Title: DPBRN Reasons for Replacement or Repair of Dental Restorations
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Heatlh Partners Research Foundation (Minnesota) (Unknown); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, University of Alabama at Birmingham
Other Study IDs: 118680; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Dental Caries
Keywords: Dental Caries; Assessments; dental materials
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to document the reasons for replacement or repair of defective restorations ("fillings") and to record the restorative material of the failed restoration and the material used in the replacement restoration on permanent ("adult") teeth.

DETAILED DESCRIPTION:
The aims of this study were to (1) quantify the prevalence of reason(s) for replacing existing restorations in DPBRN practices; (2) quantify the percentages and types of restorative materials of failed restorations that are being replaced in DPBRN practices; (3) quantify the percentages and types of restorative materials used to replace or repair failed restorations in DPBRN practices; and (4) test the hypothesis that DPBRN practitioner-investigators who reported in a previous study that they treat enamel lesions operatively are more likely in actual patients as in this study to replace entire restorations rather than do repairs and are more likely to report the clinical diagnosis of secondary caries as a reason for replacement.

ELIGIBILITY:
Inclusion Criteria:

* participants directly involved in this study were patients who sought dental treatment in the practitioner-investigators practices
* any tooth surface that was previously restored was eligible for this study, provided that it was on a permanent ("adult") tooth. This means that permanent first molars were eligible, which typically erupt at about age 6 years. This means that persons age 6 and older were enrolled in the study and there was no upper age limit.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practitioner investigators must have been enrolled in the DPBRN, completed the "Assessment of caries diagnosis & caries treatment" study; and do at least some restorative dentistry in their practices. The human subjects directly involved in this study were patients who had sought dental treatment in the DPBRN practitoners' practices.
Sampling Method: Probability Sample
Enrollment: 6368 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria V Gordan, DDS, MS, MSCI, Principal Investigator — Dental Practice-Based Research Network; Gregg H Gilbert, DDS, MBA, Study Chair — Dental Practice-Based Research Network
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org